CLINICAL TRIAL: NCT00852644
Title: Feasibility and Outcome of Cyberknife® Precision Hypofractionated Radiosurgery for the Curative Management of Non-Small Cell Lung Cancer
Brief Title: Stereotactic Radiosurgery in Treating Patients With Stage I or Stage II Non-Small Cell Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor accrual
Sponsor: Boston Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Minh Tam Truong, Chair and Associate Professor, Radiation Oncology, Boston Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-26701; CDR0000635119 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Fluorodeoxyglucose F18; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Participants to receive Cyberknife radiation therapy in 4 doses over two weeks. Dose will be determined using a dose-escalation plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- 56 Gray (LESS than 3 centimeter cohort) (Experimental): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks - 56 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
  Interventions: Procedure: computed tomography; Radiation: fludeoxyglucose F 18; Radiation: hypofractionated radiation therapy; Radiation: stereotactic radiosurgery
- 62 Gray (LESS than 3 centimeter cohort) (Experimental): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks - 62 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
  Interventions: Procedure: computed tomography; Radiation: fludeoxyglucose F 18; Radiation: hypofractionated radiation therapy; Radiation: stereotactic radiosurgery
- 68 Gray (LESS than 3 centimeter cohort) (Experimental): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks - 68 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
  Interventions: Procedure: computed tomography; Radiation: fludeoxyglucose F 18; Radiation: hypofractionated radiation therapy; Radiation: stereotactic radiosurgery
- 56 Gray (MORE than 3 centimeter cohort) (Experimental): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks - 56 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
  Interventions: Procedure: computed tomography; Radiation: fludeoxyglucose F 18; Radiation: hypofractionated radiation therapy; Radiation: stereotactic radiosurgery
- 62 Gray (MORE than 3 centimeter cohort) (Experimental): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks - 62 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
  Interventions: Procedure: computed tomography; Radiation: fludeoxyglucose F 18; Radiation: hypofractionated radiation therapy; Radiation: stereotactic radiosurgery
- 68 Gray (MORE than 3 centimeter cohort) (Experimental): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks - 68 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
  Interventions: Procedure: computed tomography; Radiation: fludeoxyglucose F 18; Radiation: hypofractionated radiation therapy; Radiation: stereotactic radiosurgery

INTERVENTIONS:
Procedure: computed tomography — Standard CT scans
Radiation: fludeoxyglucose F 18 — standard doses with CT scans
Radiation: hypofractionated radiation therapy — 4 doses over 2 weeks
Radiation: stereotactic radiosurgery — CyberKnife radiosurgery

SUMMARY:
RATIONALE: Stereotactic radiosurgery can send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of stereotactic radiosurgery in treating patients with stage I or stage II non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish the maximum tolerated dose of CyberKnife® hypofractionated stereotactic radiosurgery in patients with medically inoperable, stage I or II non-small cell lung cancer.
* To establish the relationship between positron emission tomography (PET) response and local control and survival using fludeoxyglucose F 18 PET/CT imaging before treatment and at 1, 3, 6, and 12 months after treatment.

OUTLINE: Patients undergo placement of 3 gold fiducial markers by CT-guidance or bronchoscopy. Patients then undergo CyberKnife® hypofractionated stereotactic radiosurgery over 45-120 minutes twice weekly for 2 weeks.

Patients undergo fludeoxyglucose F 18 PET/CT scan at baseline and at 1, 3, 6, and 12 months after completion of treatment.

After completion of study treatment, patients are followed periodically for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Stage I or II disease (T1-3, N0, M0)

    * T2 or T3 tumor ≤ 5 cm
    * No T3 tumors involving the central chest or mediastinum (only chest wall involvement allowed)
* Tumor deemed technically resectable, in the opinion of an experienced thoracic surgeon, AND patient deemed "medically inoperable"

  * Patients with fluorodeoxyglucose (FDG)-avidity in mediastinal lymph nodes are eligible provided they are able to undergo mediastinoscopy to confirm N0 status

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment

Exclusion Criteria:

* No history of contrast allergy
* No psychological issues that would preclude the completion of study treatment

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy or chemotherapy
* No suspected nodal metastasis that cannot be falsified by mediastinoscopy (i.e., hilar or mediastinal nodes that are either fludeoxyglucose F 18 [FDG]-avid or measure > 1 cm in short axis diameter on CT scan)
* No tumor within or touching the proximal bronchial tree, defined as a volume of 2 cm in all directions around the proximal bronchial tree (carina, right and left main stem bronchi, right and left upper lobe bronchi, bronchus intermedius, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minh Tam Truong, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Cancer Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 patients were enrolled onto this study between January 2009 and August 2012 in the Radiation Oncology Clinic at Boston Medical Center
Groups:
- 56 Gray (LESS Than 3 Centimeter Cohort); 56 Gray (MORE Than 3 Centimeter Cohort): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks at 56 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
- 62 Gray (LESS Than 3 Centimeter Cohort): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks at 62 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
- 68 Gray (LESS Than 3 Centimeter Cohort); 68 Gray (MORE Than 3 Centimeter Cohort): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks at 68 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
- 62 Gray (MORE Than 3 Centimeter Cohort): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks a 62 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
Period: Overall Study
Arm/Group | 56 Gray (LESS Than 3 Centimeter Cohort) | 62 Gray (LESS Than 3 Centimeter Cohort) | 68 Gray (LESS Than 3 Centimeter Cohort) | 56 Gray (MORE Than 3 Centimeter Cohort) | 62 Gray (MORE Than 3 Centimeter Cohort) | 68 Gray (MORE Than 3 Centimeter Cohort)
Started | 3 | 3 | 0 | 3 | 0 | 0
Completed | 3 | 3 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CyberKnife: Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
Arm/Group | CyberKnife
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Did Not Experience a Dose Limiting Toxicity in the Less Than 3 Centimeter Cohort
Description: Number of Participants Who Did Not Experience a Dose Limiting Toxicity in the less than 3 centimeter cohort
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 56 Gray (LESS Than 3 Centimeter Cohort): Dose 1 (56 gray), less than 3 centimeter cohort
- 62 Gray (LESS Less Than 3 Centimeter Cohort): Dose 2 (62 gray), less than 3 centimeter cohort
- 68 Gray (LESS Than 3 Centimeter Cohort): Dose 3 (68 gray), less than 3 centimeter cohort
Arm/Group | 56 Gray (LESS Than 3 Centimeter Cohort) | 62 Gray (LESS Less Than 3 Centimeter Cohort) | 68 Gray (LESS Than 3 Centimeter Cohort)
Number analyzed (Participants) | 3 | 3 | 0
Participants | 3 | 3 | 0

2. Primary Outcome: Maximum Tolerated Dose in the Less Than 3 Centimeter Cohort
Description: The highest tolerable dose between 56 gray, 62 gray and 68 gray has not been established as the protocol was terminated early.
Time Frame: 6 weeks
Population: The highest tolerable dose between 56 gray, 62 gray and 68 gray has not been established as the protocol was terminated early.
Units Other Than Participants: dose
Arm/Group | 56 Gray (LESS Than 3 Centimeter Cohort) | 62 Gray (LESS Less Than 3 Centimeter Cohort) | 68 Gray (LESS Than 3 Centimeter Cohort)
Number analyzed (Participants) | 0 | 0 | 0
Number analyzed (dose) | 0 | 0 | 0

3. Primary Outcome: Participants Who Did Not Experience a Dose Limiting Toxicity in the More Than 3 Centimeter Cohort
Description: The number of participants that did not experience a dose-limiting toxicity in the greater than 3 centimeter cohort
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 56 Gray (MORE Than 3 Centimeter Cohort): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks - 56 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
  computed tomography: Standard CT scans
  fludeoxyglucose F 18: standard doses with CT scans
  hypofractionated radiation therapy: 4 doses over 2 weeks
  stereotactic radiosurgery: CyberKnife radiosurgery
- 62 Gray (MORE Than 3 Centimeter Cohort): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks - 62 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
  computed tomography: Standard CT scans
  fludeoxyglucose F 18: standard doses with CT scans
  hypofractionated radiation therapy: 4 doses over 2 weeks
  stereotactic radiosurgery: CyberKnife radiosurgery
- 68 Gray (MORE Than 3 Centimeter Cohort): Intervention:
  Procedure/Surgery: computed tomography Standard CT scans
  Intervention:
  Radiation: fludeoxyglucose F 18 standard doses with CT scans
  Radiation: hypofractionated radiation therapy 4 doses over 2 weeks - 68 Gray
  Radiation: stereotactic radiosurgery CyberKnife radiosurgery
  computed tomography: Standard CT scans
  fludeoxyglucose F 18: standard doses with CT scans
  hypofractionated radiation therapy: 4 doses over 2 weeks
  stereotactic radiosurgery: CyberKnife radiosurgery
Arm/Group | 56 Gray (MORE Than 3 Centimeter Cohort) | 62 Gray (MORE Than 3 Centimeter Cohort) | 68 Gray (MORE Than 3 Centimeter Cohort)
Number analyzed (Participants) | 3 | 0 | 0
Participants | 3 | 0 | 0

4. Primary Outcome: Maximum Tolerated Dose - More Than 3 Centimeter Cohort.
Description: as for outcome 2
Time Frame: 6 weeks
Population: as for outcome 2
Units Other Than Participants: dose
Arm/Group | 56 Gray (MORE Than 3 Centimeter Cohort) | 62 Gray (MORE Than 3 Centimeter Cohort) | 68 Gray (MORE Than 3 Centimeter Cohort)
Number analyzed (Participants) | 0 | 0 | 0
Number analyzed (dose) | 0 | 0 | 0

5. Secondary Outcome: Relationship Between Positron Emission Tomography (PET) Response and Local Control and Survival
Description: Relationship between positron emission tomography (PET) response and local control and survival as measured by fludeoxyglucose F 18 PET/CT imaging
Time Frame: before treatment and at 1, 3, 6, and 12 months after treatment
Population: Data were not collected and the outcome measure was not analyzed
Arm/Group | CyberKnife
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 56 Gray (LESS Than 3 Centimeter Cohort) | 62 Gray (LESS Than 3 Centimeter Cohort) | 68 Gray (LESS Than 3 Centimeter Cohort) | 56 Gray (MORE Than 3 Centimeter Cohort) | 62 Gray (MORE Than 3 Centimeter Cohort) | 68 Gray (MORE Than 3 Centimeter Cohort)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/0 | 0/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 0/0 | 1/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 0/0 | 3/3 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 56 Gray (LESS Than 3 Centimeter Cohort) (N=3) | 62 Gray (LESS Than 3 Centimeter Cohort) (N=3) | 68 Gray (LESS Than 3 Centimeter Cohort) (N=0) | 56 Gray (MORE Than 3 Centimeter Cohort) (N=3) | 62 Gray (MORE Than 3 Centimeter Cohort) (N=0) | 68 Gray (MORE Than 3 Centimeter Cohort) (N=0)
Forced Expiratory Volume in One Second (FEV1) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
diabetes (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffusing capacity of the lungs for carbon monoxide (DLCO) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gait/walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hyperglycemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 56 Gray (LESS Than 3 Centimeter Cohort) (N=3) | 62 Gray (LESS Than 3 Centimeter Cohort) (N=3) | 68 Gray (LESS Than 3 Centimeter Cohort) (N=0) | 56 Gray (MORE Than 3 Centimeter Cohort) (N=3) | 62 Gray (MORE Than 3 Centimeter Cohort) (N=0) | 68 Gray (MORE Than 3 Centimeter Cohort) (N=0)
dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gait/walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Presented to Emergency Department with chest pain. Treated for non-ST segment elevation myocardial infarction) - Grade 1
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
heartburn (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
infection-other (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
insomnia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
musculoskeletal-other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — left sided muscle soreness
nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pulmonary fibrosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
voice changes (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The highest tolerable dose was not established in either cohort due to early termination. There were no dose limiting toxicities experienced at 56 or 62 gray (less than 3 centimeters) or 56 gray (more than 3 centimeters) at the time of study closure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes